CLINICAL TRIAL: NCT07353593
Title: Effect of Kinesio Tape Versus Systemic Dexamethasone on Postsurgical Sequels Following Extraction of Impacted Mandibular Third Molars
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ashraf elanzy (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Ashraf elanzy, Principal Investigator, Department of Oral and Maxillofacial Surgery, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M0208023os
Record Dates: First submitted 2025-12-24; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Impacted Mandibular Third Molar Extraction
Keywords: Kinesio Tape, Dexamethasone, Mandibular Third Molar, Oral Surgery, Postoperative Edema, Pain Management, Trismus, Non-Pharmacological Therapy
MeSH Terms: conditions — Agnosia; Trismus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Tape (Experimental)
  Interventions: Other: Kinesio Tape application
- Dexamethasone (Active Comparator)
  Interventions: Drug: Intramuscular Injection of Dexamethasone
- Control (Active Comparator)
  Interventions: Other: control

INTERVENTIONS:
Other: Kinesio Tape application — Kinesio Tape application after horizontal impacted mandibular third molar extraction
  Arms: Kinesio Tape
Drug: Intramuscular Injection of Dexamethasone — 8 M.g Intramuscular Injection of Dexamethasone** after horizontal impacted mandibular third molar extraction
  Arms: Dexamethasone
Other: control — left to heal without use of Dexamethasone nor Kinesio Tape after horizontal impacted mandibular third molar extraction
  Arms: Control

SUMMARY:
The surgical removal of lower wisdom teeth is a common procedure that can cause pain, facial swelling, and difficulty in opening the mouth after surgery. These symptoms are usually managed with medications such as dexamethasone, which helps reduce inflammation but may have unwanted side effects in some patients.

This study compares the use of dexamethasone with Kinesio Tape, a non-drug treatment applied to the skin, to evaluate their effectiveness in reducing pain, swelling, and limited mouth opening after wisdom tooth removal. The findings of this study may help determine whether Kinesio Tape can be a safe and effective alternative to medication for improving recovery after surgery.

DETAILED DESCRIPTION:
The extraction of impacted mandibular third molars is one of the most common procedures performed in oral and maxillofacial surgery. Despite being a routine intervention, it is frequently associated with significant postoperative complications, including pain, edema, and trismus, all of which negatively impact patient recovery and quality of life. These sequelae result from the inflammatory response induced by surgical trauma, leading to increased vascular permeability, extracellular fluid accumulation, and the release of inflammatory mediators. Given these concerns, optimizing postoperative management strategies is critical to improving patient outcomes and enhancing recovery. Traditional pharmacological interventions, particularly dexamethasone, have been widely employed due to their potent anti-inflammatory effects. However, concerns regarding systemic side effects, contraindications, and long-term implications have led to increasing interest in non-pharmacological alternatives such as Kinesio Tape (KT).

The physiological response following third molar extraction is driven by a complex interplay of cellular and molecular mechanisms aimed at tissue healing and immune regulation. Surgical trauma triggers the activation of pro-inflammatory cytokines, including tumor necrosis factor-alpha, interleukin-1 beta, and interleukin-6, which contribute to increased vascular permeability, edema formation, and nociceptor sensitization. This inflammatory cascade ultimately results in pain, swelling, and limited mouth opening due to spasm and fibrosis of the masticatory muscles, particularly the masseter and pterygoid muscles. The peak of these complications typically occurs within 48 hours postoperatively and, if not adequately managed, may lead to prolonged recovery, reduced oral function, and impaired patient satisfaction.

Dexamethasone is a long-acting glucocorticoid that exerts its effects by inhibiting the transcription of pro-inflammatory genes, thereby reducing cytokine release, stabilizing cell membranes, and preventing fluid extravasation into surrounding tissues. Evidence has shown that a single preoperative dose of dexamethasone administered via submucosal or intramuscular injection can effectively reduce postoperative swelling, trismus, and pain intensity, making it a widely adopted intervention in oral surgery. Nevertheless, despite its efficacy, systemic corticosteroids are associated with potential risks, including immunosuppression, delayed wound healing, alterations in glucose metabolism, and adrenal suppression with prolonged use. These concerns have necessitated the exploration of alternative strategies capable of achieving comparable anti-inflammatory effects without systemic exposure.

Kinesio Tape has gained increasing attention in rehabilitation medicine and sports therapy, with growing interest in its role in postoperative recovery. Designed to lift the skin, decompress underlying tissues, and enhance lymphatic drainage, KT has been proposed as an effective method for reducing edema, improving blood circulation, and modulating neuromuscular function. Unlike corticosteroids, which act at the molecular level to suppress inflammation, KT exerts its effects mechanically by redistributing interstitial pressure, facilitating fluid dynamics, and promoting natural healing mechanisms.

Clinical investigations have assessed the efficacy of KT in reducing postoperative complications following third molar extraction. Application of KT has been associated with reductions in swelling, pain intensity, and trismus during the early postoperative period, suggesting a sustained benefit in controlling tissue inflammation. Moreover, KT does not induce systemic effects, making it an attractive option for patients with contraindications to corticosteroid therapy.

Comparative evaluations between dexamethasone and KT in managing postoperative sequelae suggest that while dexamethasone provides a more immediate reduction in inflammation, KT offers a gradual and sustained improvement in edema resolution. KT application has also been associated with improved patient-reported comfort, potentially due to its continuous therapeutic effect throughout the postoperative period, in contrast to the transient pharmacological action of corticosteroids.

Despite promising findings regarding KT as an alternative or adjunct to dexamethasone, gaps remain in understanding its optimal clinical application, efficacy across diverse patient populations, and potential synergistic effects when combined with pharmacological interventions. This study aims to address these gaps by conducting a comprehensive comparative analysis of Kinesio Tape versus dexamethasone in mitigating postoperative pain, swelling, and trismus following mandibular third molar extraction. Through this investigation, the study seeks to contribute meaningful insights into the development of multimodal, minimally invasive postoperative management strategies in oral surgery.

ELIGIBILITY:
Inclusion criteria:

1. Patients (male and female) with age 20-40 years old.
2. Co-operative patients.
3. An impacted lower wisdom tooth diagnosed with a moderate to severe difficulty index according to Pell and Gregory or Pederson scale classification.104
4. Medically Free from any systemic conditions.

Exclusion criteria:

1. Uncooperative patients.
2. Smoker patients.
3. Pregnant or lactating women.
4. Women taking oral contraceptives.
5. Patient with systemic diseases.
6. Patients misunderstanding the clinical procedures of the study.
7. Individuals allergic or intolerant to Dexamethasone used in the study.
8. Patients on oral anticoagulants.
9. Uncontrolled diabetic patients.
10. Individuals with periodontal disease or active infection at the site of impacted tooth.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Facial swelling (edema) measured in millimeters at three facial points after mandibular third molar extraction | Immediately after extraction, Day 3, and Day 7 postoperatively
  Edema will be assessed using a flexible ruler at three standardized points:
  1. Lateral corner of the eye to angle of the mandible
  2. Tragus to corner of the mouth
  3. Inferior point of the angle of the mandible to lateral point of the lip commissure Measurements will be performed immediately after extraction, at 3 days, and at 7 days postoperatively.
Maximum interincisal distance (mm) to assess mouth opening after mandibular third molar extraction | Immediately after extraction, Day 3, and Day 7 postoperatively
  Mouth opening will be measured as the maximum interincisal distance using a caliper. Measurements will be taken immediately after extraction, at 3 days, and at 7 days postoperatively.
Pain intensity score after mandibular third molar extraction measured using the Visual Analog Scale (VAS, 1-10) | Immediately after extraction, Day 3, and Day 7 postoperatively
  Pain intensity will be self-reported by each participant using the Visual Analog Scale (VAS) ranging from 1 (no pain) to 10 (worst pain imaginable). Pain will be assessed immediately post-extraction, at 3 days, and at 7 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelmonem Tawfik, Prof, Principal Investigator — Mansoura University; Fakhreldin Hassan Abdelrahman, PHD, Principal Investigator — Mansoura University
Locations (1):
- Mansura Universtiy, Al Mansurah, Mansura, Egypt

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data (IPD) outside the primary research group due to the small sample size and to protect participant confidentiality.